CLINICAL TRIAL: NCT01612481
Title: Phase II Study Evaluating Strategies of Lung Surveillance of Patients Operated of High Grade Soft Tissue Sarcoma: Chest Radiograph Versus Chest CT
Brief Title: Phase II Study Evaluating Strategies of Lung Surveillance of Patients Operated of High Grade Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CASSANDRE - 1108
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Soft Tissue Sarcoma; Lung Metastasis
Keywords: soft tissue sarcoma; lung metastasis; surveillance
MeSH Terms: conditions — Sarcoma | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chest radiography (Active Comparator): clinical exam + chest radiography every 3 months during 2 years and every 6 months during 1 year
  Interventions: Procedure: chest radiography
- chest CT (Active Comparator): clinical exam + Chest CT every 3 months during 2 years and every 6 months during 1 year
  Interventions: Procedure: chest CT

INTERVENTIONS:
Procedure: chest radiography — surveillance by radiography of chest every 3 months the first 2 years then every 6 month the third, forth and fifth years
  Arms: chest radiography
Procedure: chest CT — surveillance by CT of chest every 3 months the first 2 years then every 6 month the third, forth and fifth years
  Arms: chest CT

SUMMARY:
Cancer surveillance has a significant cost and generate anxiety for the patient.

It is important to avoid exams that will not modify health support or whose results wont allow to decide.

DETAILED DESCRIPTION:
Cancer surveillance has a significant cost and generate anxiety for the patient.

It is important to avoid exams that will not modify health support or whose results wont allow to decide.

Our study will help rationalise surveillance of soft tissue sarcoma and standardize medical practices.

ELIGIBILITY:
Inclusion Criteria:

* soft tissue sarcoma, histologically proven
* tumor size > 5 cm (SBR grade 2) or whatever size (SBR grade 3)
* complete excision (R0 or R1)
* no metastasis (checked by spiral chest CT)
* social security covered
* informed signed consent

Exclusion Criteria:

* bone, visceral, uterine, retroperitoneal sarcoma
* GIST
* other malignant tumor
* patients over 70, or for whom thoracic surgery is excluded
* pneumoconiosis or known system disease
* breast feeding or pregnant woman
* patient unable to undergo trail medical follow up for geographic, social or psychological reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
proportion of patients having an isolated and operable pulmonary relapse | 2 years
  % of patients having resectable or resected lung metastasis after 2 years of surveillance

SECONDARY OUTCOMES:
evaluate quality of life | every 3 months for 2 years then every 6 months for the 3rd year
  questionnaire STAI
evaluate free disease survival | 5 years
  Time between date of inclusion and date of clinical or radiological progression
evaluate overall survival | 5 years
  time between date of inclusion and date of death (whatever the cause is)
evaluate irradiation received | 2 years
  measure of PDL (product dose length) for chest CT measure of PDS (product dose surface) for chest radiograph
estimate false positive rate | 2 years
  patients operated for non metastatic lesions patients monitored for non metastatic nodules
evaluate global health | every 3 months for 2 years then every 6 months for the 3rd year
  using scale of pain EVA
medico economic evaluation | 5 years
  sum of direct and indirect costs

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, MD, Principal Investigator — Oscar Lambret Center
Locations (3):
- France (3):
  - Centre Georges François Leclerc, Dijon
  - Oscar Lambret Center, Lille
  - Léon BERARD Center, Lyon

IPD SHARING:
Plan to Share IPD: No